

# STATISTICAL ANALYSIS PLAN

A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Phase 3 Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solutions (0.25% and 0.5%) Compared to Vehicle in the Conjunctival Allergen Challenge (Ora-CAC®) Model of Acute Allergic Conjunctivitis



Sponsor: Aldeyra Therapeutics, Inc.

131 Hartwell Ave. Lexington, MA 02421

Protocol Number: ADX-102-AC-008

Author:



Date: 20FEB2019

Version: 1.0



A Multi-Center, Double-Masked, Randomized, Parallel-Group, Vehicle-Controlled, Phase 3 Clinical Trial to Assess the Safety and Efficacy of Reproxalap Ophthalmic Solutions (0.25% and 0.5%) Compared to Vehicle in the Conjunctival Allergen Challenge (Ora-CAC®) Model of Acute Allergic Conjunctivitis

Protocol Number:

ADX-102-AC-008

Version:

1.0

Date:

20FEB2019

Statistical Analysis Plan Approval

| _ | 40 | KOVEX |
|--------------|----|-------|
| Prepared by: | | |
| N. | | |
| Reviewed by: | | |
| 9 | | |
| Approved by: | | |
| Approved by: | | |

# Protocol ADX-102-AC-008 SAP, Version 1.0



#### **Table of Contents**

| 1. | Introduction | 6 |
|------|--------------------------------------------------|----|
| 2. | Study Objectives | 6 |
| 3. | Study Design and Procedures | 6 |
| 3.1 | General Study Design | 6 |
| 3.2 | Schedule of Visits and Assessments | 7 |
| 4. | Study Endpoints | 8 |
| 4.1 | Primary Efficacy Endpoints | 8 |
| 4.2 | Key Secondary Efficacy Endpoint | 8 |
| 4.3 | Additional Secondary Efficacy Variables | 8 |
| 4.4 | Safety Variables | 8 |
| 4.5 | Statistical Hypotheses | 9 |
| 5. | Study Treatments | 9 |
| 5.1 | Method of Assigning Subjects to Treatment Groups | 10 |
| 5.2 | Masking and Unmasking | 10 |
| 6. | Sample Size and Power Considerations | 10 |
| 7. | Data Preparation | 11 |
| 8. | Analysis Populations | 12 |
| 8.1 | Intent-to-Treat | 12 |
| 8.2 | Per-Protocol | 12 |
| 8.3 | Safety | 12 |
| 9. | General Statistical Considerations | 12 |
| 9.1 | Unit of Analysis | 12 |
| 9.2 | Missing or Inconclusive Data Handling | 12 |
| 9.3 | Definition of Baseline | 14 |
| 9.4 | Data Analysis Conventions | 14 |
| 9.5 | Adjustments for Multiplicity | 15 |
| 10. | Disposition of Subjects | 15 |
| 11. | Demographic and Pretreatment Variables | 16 |
| 11.1 | Demographic Variables | 16 |
| 11.2 | Pretreatment Variables | 16 |
| 12. | Medical History and Concomitant Medications | 17 |
| 12.1 | Medical History | 17 |
| 12.2 | 2 Concomitant Medications | 17 |
| 13. | Exposure to Investigational Product | 17 |

# Protocol ADX-102-AC-008 SAP, Version 1.0



| 14. | Efficacy Analyses1 | 8 |
|------|-----------------------------------------|---|
| 14.1 | Primary Analysis1 | 8 |
| 14.2 | Secondary Analyses1 | 9 |
| 14 | 2.1 Ocular Itching Responders Analysis1 | 9 |
| 14 | 2.2 Time to Response2 | 1 |
| 14 | 2.3 Ocular Itching2 | 2 |
| 15. | Safety Analyses2 | 3 |
| 15.1 | Adverse Events/Adverse Drug Reactions2 | 4 |
| 15.2 | Visual Acuity2 | 5 |
| 15.3 | Slit-Lamp Biomicroscopy Examination2 | 5 |
| 15.4 | Intraocular Pressure2 | 6 |
| 15.5 | Dilated Fundoscopy Examination2 | 6 |
| 15.6 | Conjunctival Redness2 | 6 |
| 16. | Interim Analyses2 | 7 |
| 17. | Changes from Protocol-Stated Analyses2 | 7 |
| 18. | Revision History2 | 7 |
| 19. | Tables2 | 7 |
| 20. | Listings2 | 9 |
| 21. | Figures | 0 |



## **List of Abbreviations**

| AE | Adverse Event |
|---|---|
| ANCOVA | Analysis of Covariance |
| ATC | Anatomical Therapeutic Chemical Classification |
| AUC <sub>t1-t2</sub> | Area Under the Curve |
| CAC | Conjunctival Allergen Challenge |
| CI | Confidence Interval |
| CS | Clinically Significant (when used in the context of safety); Compound Symmetric (when used in the context of covariance structures) |
| eCRF | Electronic Case Report Form |
| ETDRS | Early Treatment of Diabetic Retinopathy Study |
| GEE | Generalized Estimating Equation |
| HIPAA | Health Information Portability and Accountability Act |
| ICH | International Conference on Harmonisation |
| IOP | Intraocular Pressure |
| IP | Investigational Product |
| ITT | Intent-to-Treat |
| LM | Linear Model |
| logMAR | Logarithm of the Minimum Angle of Resolution |
| LS | Least Squares |
| MCMC | Markov Chain Monte Carlo |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NA | Not Applicable |
| NCS | Not Clinically Significant |
| OD | Right Eye |
| OS | Left Eye |
| PDF | Portable Document Format |
| PP | Per Protocol |
| PT | Preferred Term |
| RTF | Rich Text Format |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Statistics and Data Corporation, Incorporated |
| SOC | System Organ Class |
| TEAE | Treatment-Emergent Adverse Event |
| VA | Visual Acuity |
| WHO DDE | World Health Organization Drug Dictionary Enhanced |



#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to describe the planned analyses and reporting for protocol ADX-102-AC-008, Version 1.0 dated 15FEB2018.

This SAP is being written with due consideration of the recommendations outlined in the most recent International Conference on Harmonisation (ICH) E9 Guideline entitled Guidance for Industry: Statistical Principles for Clinical Trials and the most recent ICH E3 Guideline, entitled Guidance for Industry: Structure and Content of Clinical Study Reports.

This SAP describes the data that will be analyzed and the subject characteristics, efficacy, and safety assessments that will be evaluated. This SAP provides details of the specific statistical methods that will be used. The statistical analysis methods presented in this document will supersede the statistical analysis methods described in the clinical protocol. If additional analyses are required to supplement the planned analyses described in this SAP, they may be completed as post-hoc analyses and will be identified as such in the clinical study report.

#### 2. Study Objectives

The objective of this study is to evaluate the safety and efficacy of Reproxalap Ophthalmic Solutions (0.25% and 0.5%) compared to Vehicle Ophthalmic Solution for the treatment of ocular itching associated with acute allergic conjunctivitis.

#### 3. Study Design and Procedures

#### 3.1 General Study Design

| This is a multi-center, double-masked, randomized, parallel-group, vehicle-controlled Phase 3 clinical |
|---|
| trial will enroll approximately to evaluate the safety and efficacy of Reproxalap Ophthalmic |
| Solutions (0.25% and 0.5%) compared to Vehicle Ophthalmic Solution for the treatment of ocular itching |
| associated with acute (seasonal) allergic conjunctivitis. |
| The trial will be comprised of |
| Subjects who meet the entry |
| criteria for itching and redness response |
| to receive bilateral administration of either Reproxalap Ophthalmic |
| Solution 0.25%, Reproxalap Ophthalmic Solution 0.5%, or Vehicle Ophthalmic Solution. |



Study visits will be referred to in all tables and listings as the visit and expected study day corresponding to the visit to enable reviewers to understand the assessment timing without referring to the protocol visit schedule. The following table shows the scheduled study visits, their planned study day (note that there is no Day 0 and that Day 1 corresponds to the day of randomization), and the acceptable visit window for each study visit:

| Scheduled Visit | Planned Study Day | Visit Window |
|-----------------|-------------------|--------------|
| Screening | Day -22 | - 39 Days |
| Visit 1 | Day -21 | ± 3 Days |
| Visit 2 | Day -14 | ± 3 Days |
| Visit 3 | Day 1 | NA |

#### 3.2 Schedule of Visits and Assessments

The schedule of visits and assessments is provided below.





| | | STATISTICS & I | DATA CORPORATION |
|---|-----------------|----------------|------------------|
| | <b>-</b> | | |
| 1 | Study Endnoints | | |

## 4. Study Endpoints

## 4.1 Primary Efficacy Endpoints

The primary efficacy endpoint is the following:

Ocular itching score

## 4.2 Key Secondary Efficacy Endpoint

The key secondary efficacy endpoint is the following:

## 4.3 Additional Secondary Efficacy Variables

The additional secondary efficacy endpoints are the following:

The time to response

Ocular itching score

#### 4.4 Safety Variables

The safety variables include the following:

#### Protocol ADX-102-AC-008 SAP, Version 1.0



- Adverse Events (AE) (reported, elicited, and observed);
- Visual Acuity (VA)



- Slit-lamp Biomicroscopy;
- Intraocular Pressure (IOP);
- Dilated Fundoscopy;
- Conjunctival Redness.

## 4.5 Statistical Hypotheses

The null and alternative hypotheses, based on the primary and key secondary efficacy endpoints, are as follows:

| _ | |
|--------------|--------------------------------|
| Γο control t | the overall Type I error rate, |
| | 71 |

#### 5. Study Treatments

The study consists of three treatment arms:

- Reproxalap Ophthalmic Solution 0.25%;
- Reproxalap Ophthalmic Solution 0.5%;



Vehicle Ophthalmic Solution.

#### 5.1 Method of Assigning Subjects to Treatment Groups

All subjects screened for the trial who sign an informed consent form will be assigned a 3-digit screening number that will be entered in the Screening and Enrollment Log. Screening numbers will be assigned in a sequential order beginning with 001. Randomization will be used to avoid bias in the assignment of subjects to treatments, to increase the likelihood that known and unknown subject attributes

Once a subject meets all qualification criteria

they will be enrolled and randomly assigned to masked treatment

Subjects will be assigned the lowest 4-digit randomization number available at the investigative site within the appropriate stratum.

#### 5.2 Masking and Unmasking

When medically necessary, the investigator may need to determine what treatment has been assigned to a subject. The investigator should make every effort to contact Ora to discuss the subject's emergency situation and the need to unmask a trial subject prior to unmasking IP.

If the investigator determines that emergency unmasking is necessary, the investigator should identify the given subject's trial drug kit, which contains a scratch-off laminate under which the treatment is identified along with the associated lot number. In order to unmask, the investigator should scratch off the laminate, using a flat object and applying pressure, to reveal the treatment assigned for that subject. The emergency unmasking should be performed by the designated site personnel. The investigator must also indicate in source documents and in the electronic case report form (eCRF) that the mask was broken and provide the date, time, and reason for breaking the mask. Any AE or serious AE (SAE) associated with breaking the mask must be recorded and reported as specified in this protocol. The investigator has the responsibility to contact Ora within 24 hours of breaking the blind.

If treatment assignment is unmasked, the IP will be discontinued immediately, and the subject will be discontinued from the trial.

## 6. Sample Size and Power Considerations



#### 7. Data Preparation

After data are entered into the clinical study database, electronic edit checks and data review will be performed. All data validation specifications and procedures are detailed in the Data Validation Manual as a separate document. When the database has been declared to be complete and accurate, the database will be locked. Any changes to the database after data have been locked can only be made with the approval of the Sponsor and Ora in consultation with SDC.

All analyses outlined in this document will be carried out after the following have occurred:

| • |
|---|



| 8. Anal | vsis Po | pulations |
|---------|---------|-----------|
|---------|---------|-----------|

8.1 Intent-to-Treat

| The Intent-to-Treat (ITT) population consists of |
|----------------------------------------------------------|
| 8.2 Per-Protocol |
| The Per-Protocol (PP) population is |
| · |
| 8.3 Safety |
| The Safety population includes |
| 9. General Statistical Considerations |
| 9.1 Unit of Analysis |
| 9.2 Missing or Inconclusive Data Handling |
| The primary analysis of ocular itching will be conducted |



# Protocol ADX-102-AC-008 SAP, Version 1.0



| The key secondary endpoint |
|---|
| will be analyzed |
| 9.3 Definition of Baseline |
| For the primary efficacy endpoin |
| When analyzing ocular itching scores |
| when analyzing occilar itching scores |
| 9.4 Data Analysis Conventions |
| Data analysis will be performed by SDC using Output will be provided in |
| rich text format (RTF) for tables and portable document format (PDF) for tables, listings, and figures |
| using landscape orientation. |



| _ |
|---------------------------------------|
| · |
| 9.5 Adjustments for Multiplicity |
| 10. Disposition of Subjects |
| Subject disposition will be presented |



| Subject listings will be provided |
|---|
| Protocol violations will be summarized |
| Totada Viciationa will be administrated |
| A subject listing will be provided |
| 11. Demographic and Pretreatment Variables |
| 11.1 Demographic Variables |
| The demographic variables collected |
| A subject listing that includes all demographic variables will be provided. |
| 11.2 Pretreatment Variables |
| will be provided in a subject listing. |



# 12. Medical History and Concomitant Medications

# 12.1 Medical History

| Medical history will be coded using Medical Dictionary for Regulatory Activities (MedDRA) 21.0. |
|---|
| Listings of medical history will be generated |
| 12.2 Concomitant Medications |
| Prior and concomitant medications will be coded using the World Health Organization Drug Dictionary |
| Listings of concomitant medications will be generated |
| separately for ocular and non-ocular data. |
| 13. Exposure to Investigational Product |
| 10. Exposure to investigational i founct |

A listing of IP instillation for all subjects will also be provided.



# 14. Efficacy Analyses 14.1 **Primary Analysis** The primary efficacy variable is ocular itching score



| STATISTICS & DATA CONTONATION |
|-------------------------------|

# 14.2 Secondary Analyses

# 14.2.1 Ocular Itching Responders Analysis

| The key secondary efficacy endpoint |
|-------------------------------------|







## 14.2.2 Time to Response





## 14.2.3 Ocular Itching





| A listing of ocular itching scores for all subjects will also be provided. 15. Safety Analyses The safety outcomes |
|---|
| The safety outcomes All safety analyses will be conducted using the Safety Population. |



### 15.1 Adverse Events/Adverse Drug Reactions

AEs, SAEs and adverse drug reactions are defined in the study protocol. All AEs will be coded using MedDRA 21.0. Treatment-emergent adverse events (TEAEs) are defined as any event that occurs or worsens on or after the day that randomized study treatment is initiated.

#### Relationship to IP

The relationship of each AE to the IP should be determined by the investigator using the following categories:

- Not related;
- Unlikely to be related;
- · Possibly related;
- Probably related;
- Definitely related.

#### Severity

Severity will be classified as mild, moderate or severe. Missing severity for AEs and TEAEs will be counted as 'Severe'.

| • | |
|---|---|
| | - |



| • | study |
|---------------------------------------------------------|-------|
| treatment discontinuation. | |
| 15.2 Visual Acuity | |
| VA will be measured | |
| Results for VA will be presented in a data listing. | |
| 15.3 Slit-Lamp Biomicroscopy Examination | |
| A slit-lamp biomicroscopy examination will be performed | |



| A subject listing of the slit-lamp biomicroscopy parameters will also be produced. |
|---|
| 15.4 Intraocular Pressure |
| IOP will be measured |
| IOP will be listed for each eye at each visit. |
| 15.5 Dilated Fundoscopy Examination Dilated fundus examinations will be performed |
| Blated fulldus examinations will be performed |
| i <b></b> |
| Results will be listed for both eyes at each visit. |
| 15.6 Conjunctival Redness |
| Conjunctival redness will be assessed |



| . Results will be listed |
|--------------------------|

#### 16. Interim Analyses

No interim analysis is planned for this study.

# 17. Changes from Protocol-Stated Analyses

## 18. Revision History

#### 19. Tables

Tables in italicized font will be produced contingent upon the amount of missing data as defined previously.

| Table Number | Title | Population |
|---|---|---|
| 14.1.1.1 | Subject Disposition | ITT Population |
| 14.1.1.2 | Protocol Violations | ITT Population |
| 14.1.2.1 | Demographics and Baseline Characteristics | ITT Population |
| 14.1.2.2 | Demographics and Baseline Characteristics | Safety Population |
| 14.1.3.1 | Ocular Medical History | ITT Population |
| 14.1.3.2 | Non-Ocular Medical History | ITT Population |
| 14.1.4.1 | Prior and Concomitant Ocular Medications by<br>Treatment Group, Drug Class and Preferred Name | ITT Population |
| 14.1.4.2 | Prior and Concomitant Non-Ocular Medications by Treatment Group, Drug Class and Preferred Name | ITT Population |
| 14.1.5 | Investigational Product Instillation | Safety Population |
| 14.2.1.1 | Summary of Ocular Itching | ITT Population with Observed Data Only |
| 14.2.1.2 | Summary of Ocular Itching | ITT Population with Multiple<br>Imputations (MCMC) |
| 14.2.1.3 | Summary of Ocular Itching | ITT Population with Multiple<br>Imputations (Control-Based<br>Pattern Mixture Model) |
| 14.2.1.4 | Summary of Ocular Itching | PP Population with Observed Data Only |
| 14.2.2.1.1 | Ocular Itching | ITT Population with Observed Data Only |
| 14.2.2.1.2 | Ocular Itching | ITT Population with Multiple<br>Imputations (MCMC) |



| Table Number | Title | Population |
|---|---|---|
| 14.2.2.1.3 | Ocular Itching | ITT Population with Multiple |
| | | Imputations (Control-Based |
| 14.2.2.2.1 | Ocular Itching | Pattern Mixture Model) ITT Population with Observed |
| 14.2.2.2.1 | Octilar riching | Data Only |
| 14.2.2.2.2 | Ocular Itching | PP Population with Observed |
| | | Data Only |
| 14.2.3.1 | Ocular Itching | ITT Population with Observed Data Only |
| 14.2.3.2 | Ocular Itching | PP Population with Observed Data Only |
| 14.2.4.1 | Ocular Itching | ITT Population with Observed Data Only |
| 14.2.4.2 | Ocular Itching | PP Population with Observed Data Only |
| 14.3.1.1 | Adverse Event Summary | Safety Population |
| 14.3.1.2 | Summary of All Ocular Adverse Events by System | Safety Population |
| | Organ Class and Preferred Term | |
| 14.3.1.3 | Summary of All Non-Ocular Adverse Events by | Safety Population |
| | System Organ Class and Preferred Term | |
| 14.3.1.4 | Summary of All Ocular Treatment-Emergent | Safety Population |
| | Adverse Events by System Organ Class and Preferred Term | |
| 14.3.1.5 | Summary of All Non-Ocular Treatment-Emergent | Safety Population |
| 1 1.5.1.5 | Adverse Events by System Organ Class and | Calciy i opalation |
| | Preferred Term | |
| 14.3.1.6 | Summary of All Ocular Treatment-Emergent | Safety Population |
| | Adverse Events Suspected to be Related to | |
| | Investigational Product by System Organ Class and Preferred Term | |
| 14.3.1.7 | Summary of All Non-Ocular Treatment-Emergent | Safety Population |
| 14.5.1.7 | Adverse Events Suspected to be Related to | Calcty i optilation |
| | Investigational Product by System Organ Class and | |
| | Preferred Term | |
| 14.3.1.8 | Summary of All Ocular Serious Adverse Events by<br>System Organ Class and Preferred Term | Safety Population |
| 14.3.1.9 | Summary of All Non-Ocular Serious Adverse | Safety Population |
| | Events by System Organ Class and Preferred Term | |
| 14.3.1.10 | Summary of All Ocular Treatment-Emergent | Safety Population |
| | Adverse Events by System Organ Class, Preferred Term, and Maximal Severity | |
| 14.3.1.11 | Summary of All Non-Ocular Treatment-Emergent | Safety Population |
| 17.0.1.11 | Adverse Events by System Organ Class, Preferred | Calcty i opulation |
| | Term, and Maximal Severity | |
| 14.3.2 | Visual Acuity | Safety Population |
| 14.3.3.1 | Slit-Lamp Biomicroscopy | Safety Population |
| 14.3.3.2 | Shift in Slit-Lamp Biomicroscopy | Safety Population |
| 14.3.4 | Intraocular Pressure | Safety Population |



| Table Number | Title | Population |
|--------------|-------------------------------------|-------------------|
| 14.3.5.1 | Dilated Fundus Examination | Safety Population |
| 14.3.5.2 | Shift in Dilated Fundus Examination | Safety Population |
| 14.3.6 | Conjunctival Redness | Safety Population |

# 20. Listings

| Listing<br>Number | Title |
|-------------------|------------------------------------------------------|
| 16.1.7 | Randomization Schedule |
| 16.2.1 | Subject Disposition |
| 16.2.2 | Protocol Violations |
| 16.2.3.1 | Study Population Inclusion |
| 16.2.3.2 | Inclusion and Exclusion Criteria |
| 16.2.4.1 | Demographics |
| 16.2.4.2 | Ocular Medical History |
| 16.2.4.3 | Non-Ocular Medical History |
| 16.2.4.4 | Prior and Concomitant Ocular Medications |
| 16.2.4.5 | Prior and Concomitant Non-Ocular Medications |
| 16.2.4.6 | Skin Test |
| 16.2.5.1 | Instillation of Investigational Product |
| 16.2.5.2 | Conjunctival Allergen Challenge |
| 16.2.5.3 | Relief Drop Instillation |
| 16.2.6 | Ocular Itching |
| 16.2.7.1 | All Adverse Events |
| 16.2.7.2 | All Serious Adverse Events |
| 16.2.7.3 | Adverse Events Leading to Death |
| 16.2.7.4 | Adverse Events Leading to Study Treatment Withdrawal |
| 16.2.8.1 | Visual Acuity |
| 16.2.8.2 | Slit-Lamp Biomicroscopy |
| 16.2.8.3 | Intraocular Pressure |
| 16.2.8.4 | Dilated Fundus Examination |
| 16.2.8.5 | Urine Pregnancy Test for Female Subjects |
| 16.2.8.6 | Conjunctival Redness |



# 21. Figures

| Figure<br>Number | Title | Population |
|---|---|---|
| 14.2.1.1 | Ocular Itching Score | ITT Population with<br>Observed Data Only |
| 14.2.1.2 | Ocular Itching Score | PP Population with<br>Observed Data Only |
| 14.2.1.3 | Ocular Itching Score | ITT Population with<br>Observed Data Only |
| 14.2.1.4 | Ocular Itching Score | PP Population with<br>Observed Data Only |